CLINICAL TRIAL: NCT05787483
Title: Evaluating Biopsychosocial Outcomes of Mindfulness-based Instruction in Adolescence
Brief Title: Biopsychosocial Outcomes of Mindfulness-based Instruction
Acronym: MindUP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Caroline G. Richter, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-300010662; UAB (Other Grant/Funding Number: UAB)
Record Dates: First submitted 2023-03-01; First posted 2023-03-28 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Specific Learning Disability; Mental Health Issue
Keywords: mindfulness-based-intervention; social and emotional learning; anxiety; stress; affect; executive function; academic achievement
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MindUP group (Experimental): Teachers in the MindUP group will deliver the program lessons twice a week for 30 minutes (1 hour per week) for 12 weeks. Based on previous studies, 12 weeks should be sufficient to cover the content from the 17 lessons.
  Interventions: Behavioral: MindUP group
- active control group (Active Comparator): business as usual; regular wellness or SEL classes
  Interventions: Behavioral: active control group

INTERVENTIONS:
Behavioral: MindUP group — MindUP is a Collaborative for Academic, Social, and Emotional Learning SELect (CASEL) program, meaning the program is evidence-based and meets the adequate criteria for developing students' social and emotional competence at the highest level. MindUP addresses all five components of the CASEL SEL Framework: self-awareness, social awareness, self-management, responsible decision-making, and relationship skills (CASEL, 2020). Students are taught how the workings of the brain are related to emotions, behaviors, decision making, and learning. MindUP is the first program to provide clear instruction in both SEL and mindfulness.
  Arms: MindUP group
Behavioral: active control group — business as usual; regular wellness or SEL classes
  Arms: active control group

SUMMARY:
Over 20% of adolescents living in the United States have a diagnosable psychiatric disorder. However, most adolescents who need mental health services do not receive them due to many reasons, including low resources in families and communities, stigma, lack of mental health providers, and other barriers to mental health care access. Alabama currently ranks 50th in access to mental healthcare and 51st (LAST) in mental healthcare provider availability with only one mental healthcare provider for every 920 persons in need. Most adolescents attend school, so delivering mental health services in the school setting eliminates many barriers to mental health care access. From the point of prevention, participation in universal social and emotional learning (SEL) programs within the school setting improves social and emotional skills, behaviors, attitudes, and academic performance. Mindfulness-based instruction is a promising approach to SEL for improving psychological functioning that is evidence-based, widely available, and scalable to various populations and settings. This project aims to investigate whether a SEL program that incorporates mindfulness-based instruction (MindUP) leads to improvements in not only self-reported well-being (i.e., anxiety, mindful attention, perceived stress, and positive and negative affect), but also objectively measured executive functioning, academic achievement, and regulation of stress physiology. The investigators will partner with schools that serve historically underserved students to test the effectiveness of the MindUP program in 5th and 6th graders. This study has the potential to benefit underserved students and their teachers who will receive training on sustainable implementation of the MindUP curriculum.

ELIGIBILITY:
Inclusion Criteria:

* Fifth grade students at i3 Academy
* fifth and sixth grade students at Tarrant Intermediate School
* 6th through 8th grade students at Spring Valley School
* All students enrolled in general education will be invited to participate in the study

Exclusion Criteria:

* those with medical, developmental, or psychiatric conditions that compromise their ability to provide valid self-reports or complete other study procedures
* only one child per family will be allowed to participate to avoid dependency in data due to clustering within families

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2023-08-14 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2024-10-16 (Actual)

PRIMARY OUTCOMES:
Anxiety - change | Five times: baseline (prior to start of the program), week 4, week 8, after the completion of the program, and a three-month follow-up
  Autonomic reactions subscale of Children's Test Anxiety Scale (CTAS): has 9-items that ask the students to respond in terms of how they think, feel, or act during a test. All the questions start with the same stem, ''While I am taking tests…'' (e.g., "I feel nervous"; "My head hurts"). Students are asked to choose between four response options (i.e., almost never, 1; some of the time, 2; most of the time, 3; almost always, 4).
Mindful attention - change | Five times: baseline (prior to start of the program), week 4, week 8, immediately after the completion of the program (week 13), and a three-month follow-up
  Mindful Attention Awareness Scale-Children (MAAS-C): has 15 items and measures the frequency of mindful states over time. Students are asked to rate how frequently they experience certain state in a 6-point Likert scale ranging from almost never to almost always (e.g., "I could be feeling a certain way and not realize it until later"; "I break or spill things because of carelessness, not paying attention, or thinking of something else").

SECONDARY OUTCOMES:
Positive and negative affect - change | 12 times - once per week
  The investigators will assess children's positive and negative affect weekly (12 times) using the Positive and Negative Affect Scale - child version. This will allow us to observe if there is change in student's affect due to the intervention. This is a 30-item scale in which the student is asked to rate in a 5-item scale ("not much or not al all" to "a lot") how much they felt certain positive and negative feelings and emotions during the past weeks (e.g., happy, sad, excited, ashamed, energetic, calm).
Stress self-report - change | Five times: baseline (prior to start of the program), week 4, week 8, immediately after the completion of the program (week 13), and a three-month follow-up
  Self-report measure of perceived stress (Perceived Stress Scale - Child, PSS-C): has 13 items and is a measure of perceived stress developed for children aged 5 to 18 years. Students are asked questions about their feelings and thoughts during the previous week (e.g., "In the last week, how often did you feel rushed or hurried?"). Items are rated on a four-point scale from "0" (Never) to "3" (Very Often).
Cortisol - change | Five times: baseline (prior to start of the program), week 4, week 8, immediately after the completion of the program (week 13), and a three-month follow-up
  Stress and inflammation biomarkers in the students' saliva: Hypothalamic-pituitary-adrenocortical (HPA) regulation and inflammation will be assessed by measuring the presence of cortisol. A sample of 1ml of saliva will be collected at each time point, three times within one day (9 A.M., 11:30 A.M., 2:30 P.M.)
Dehydroepiandrosterone (DHEA) - change | Five times: baseline (prior to start of the program), week 4, week 8, immediately after the completion of the program (week 13), and a three-month follow-up
  Stress and inflammation biomarkers in the students' saliva: Hypothalamic-pituitary-adrenocortical (HPA) regulation and inflammation will be assessed by measuring the presence of DHEA. A sample of 1ml of saliva will be collected at each time point, three times within one day (9 A.M., 11:30 A.M., 2:30 P.M.)
C-reactive protein (CRP) - change | Five times: baseline (prior to start of the program), week 4, week 8, immediately after the completion of the program (week 13), and a three-month follow-up
  Stress and inflammation biomarkers in the students' saliva: Hypothalamic-pituitary-adrenocortical (HPA) regulation and inflammation will be assessed by measuring the presence of CRP. A sample of 1ml of saliva will be collected at each time point, three times within one day (9 A.M., 11:30 A.M., 2:30 P.M.)

OTHER OUTCOMES:
Executive function: Flanker Inhibitory Control & Attention Test (Flanker) - change | Five times: baseline (prior to start of the program), week 4, week 8, immediately after the completion of the program (week 13), and a three-month follow-up
  The Flanker task from the NIH Toolbox Cognition Battery measures the child's ability to inhibit visual attention to irrelevant dimensions. The scoring procedure integrates both accuracy and reaction time. T-scores based on the participant's chronological age will be computed. T-scores range from 20 to 80 and have a mean of 50 and a standard deviation of 10. Higher scores mean a better outcome. The average time to complete the task is 4 minutes.
Executive function: Dimensional Change Card Sort Test (DCCS) - change | Five times: baseline (prior to start of the program), week 4, week 8, immediately after the completion of the program (week 13), and a three-month follow-up
  The DCCS from the NIH Toolbox Cognition Battery measures the child's ability to shift from one rule to another (the child is asked to match an object with another based on shape and then based on color). The scoring procedure integrates both accuracy and reaction time. T-scores based on the participant's chronological age will be computed. T-scores range from 20 to 80 and have a mean of 50 and a standard deviation of 10. Higher scores mean a better outcome. The average time to complete the task is 4 minutes.
Behavior Regulation - change | Five times: baseline (prior to start of the program), week 4, week 8, immediately after the completion of the program (week 13), and a three-month follow-up
  Teachers who are not responsible for teaching either group (MindUP or control) will complete the Behavior Regulation Index (BRI, 13 items) of the Behavior Rating Inventory of Executive Function (BRIEF), an ecologically valid measure of school-related executive performance. Teachers should take five minutes to complete these items per child. T-scores will be computed based on the child's chronological age. T-scores at or below 59 are considered to be within the typical range. T-scores of 60-64 are in the mildly elevated range, and scores equal to or exceeding 65 are considered to be significantly elevated. Thus, higher scores mean a worse outcome.
Emotion Regulation - change | Five times: baseline (prior to start of the program), week 4, week 8, immediately after the completion of the program (week 13), and a three-month follow-up
  Teachers who are not responsible for teaching either group (MindUP or control) will complete the Emotion Regulation Index (ERI, 16 items) of the Behavior Rating Inventory of Executive Function (BRIEF), an ecologically valid measure of school-related executive performance. Teachers should take five minutes to complete these items per child. T-scores will be computed based on the child's chronological age. T-scores at or below 59 are considered to be within the typical range. T-scores of 60-64 are in the mildly elevated range, and scores equal to or exceeding 65 are considered to be significantly elevated. Thus, higher scores mean a worse outcome.
Academic achievement - change | Five times: baseline (prior to start of the program), week 4, week 8, immediately after the completion of the program (week 13), and a three-month follow-up
  To measure academic achievement, children will complete two subtests of the Woodcock-Johnson-IV: Passage Comprehension and Calculation. In the Passage Comprehension subtest, the child is asked to determine a missing key word in a written passage. In the Calculation subtest, children are asked to complete a series of arithmetic problems arranged in order of difficulty (e.g., 5 + 2 = ?; 42 +21 +13 = ?). Children should take five minutes to complete each of the subtests. All of these five measures are standardized and provide age-corrected standard scores, for which the normative mean is 100 and the standard deviation is 15.

CONTACTS AND LOCATIONS:
Locations (1):
- Spring Valley School, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Belliveau C, Nagy C, Escobar S, Mechawar N, Turecki G, Rej S, Torres-Platas SG. Effects of Mindfulness-Based Cognitive Therapy on Peripheral Markers of Stress and Inflammation in Older-Adults With Depression and Anxiety: A Parallel Analysis of a Randomized Controlled Trial. Front Psychiatry. 2021 Dec 24;12:804269. doi: 10.3389/fpsyt.2021.804269. eCollection 2021. PMID 35002817
- [Background] Cummings JR, Ponce NA, Mays VM. Comparing racial/ethnic differences in mental health service use among high-need subpopulations across clinical and school-based settings. J Adolesc Health. 2010 Jun;46(6):603-6. doi: 10.1016/j.jadohealth.2009.11.221. Epub 2010 Feb 4. PMID 20472219
- [Background] Dunning DL, Griffiths K, Kuyken W, Crane C, Foulkes L, Parker J, Dalgleish T. Research Review: The effects of mindfulness-based interventions on cognition and mental health in children and adolescents - a meta-analysis of randomized controlled trials. J Child Psychol Psychiatry. 2019 Mar;60(3):244-258. doi: 10.1111/jcpp.12980. Epub 2018 Oct 22. PMID 30345511
- [Background] Schonert-Reichl KA, Oberle E, Lawlor MS, Abbott D, Thomson K, Oberlander TF, Diamond A. Enhancing cognitive and social-emotional development through a simple-to-administer mindfulness-based school program for elementary school children: a randomized controlled trial. Dev Psychol. 2015 Jan;51(1):52-66. doi: 10.1037/a0038454. PMID 25546595
- [Background] Morganti A, Ambrosi B, Sala C, Cianci L, Bochicchio D, Turolo L, Zanchetti A. Effects of angiotensin II blockade on the responses of the pituitary-adrenal axis to corticotropin-releasing factor in humans. J Cardiovasc Pharmacol. 1987;10 Suppl 7:S167-9. doi: 10.1097/00005344-198706107-00038. PMID 2485058
- [Background] Wren, D. G., & Benson, J. (2004). Measuring test anxiety in children: Scale development and internal construct validation. Anxiety, Stress & Coping, 17(3), 227-240. https://doi.org/10.1080/10615800412331292606
- [Background] Lawlor, M. S., Schonert-Reichl, K. A., Gadermann, A. M., & Zumbo, B. D. (2014). A validation study of the mindful attention awareness scale adapted for children. Mindfulness, 5(6), 730-741. https://doi.org/10.1007/s12671-013-0228-4
- [Background] Laurent, J., Catanzaro, S. J., Joiner Jr., T. E., Rudolph, K. D., Potter, K. I., Lambert, S., Osborne, L., & Gathright, T. (1999). A measure of positive and negative affect for children: Scale development and preliminary validation. Psychological Assessment, 11(3), 326-338. https://doi.org/10.1037/1040-3590.11.3.326
- [Background] White, B. P., & White, B. P. (2014). The perceived stress scale for children: A pilot study in a sample of 153 children. International Journal of Pediatrics and Child Health, 2(2), 45-52. https://doi.org/10.12974/2311-8687.2014.02.02.4
- [Background] Gioia, G. A., Isquith, P. K., Guy, S. C., & Kenworthy, L. (2015). BRIEF-2: Behavior rating inventory of executive function: Professional manual. Psychological Assessment Resources.
- [Background] Weintraub S, Dikmen SS, Heaton RK, Tulsky DS, Zelazo PD, Bauer PJ, Carlozzi NE, Slotkin J, Blitz D, Wallner-Allen K, Fox NA, Beaumont JL, Mungas D, Nowinski CJ, Richler J, Deocampo JA, Anderson JE, Manly JJ, Borosh B, Havlik R, Conway K, Edwards E, Freund L, King JW, Moy C, Witt E, Gershon RC. Cognition assessment using the NIH Toolbox. Neurology. 2013 Mar 12;80(11 Suppl 3):S54-64. doi: 10.1212/WNL.0b013e3182872ded. PMID 23479546
- [Background] Rueda MR, Fan J, McCandliss BD, Halparin JD, Gruber DB, Lercari LP, Posner MI. Development of attentional networks in childhood. Neuropsychologia. 2004;42(8):1029-40. doi: 10.1016/j.neuropsychologia.2003.12.012. PMID 15093142
- [Background] Zelazo PD. The Dimensional Change Card Sort (DCCS): a method of assessing executive function in children. Nat Protoc. 2006;1(1):297-301. doi: 10.1038/nprot.2006.46. PMID 17406248
- [Background] Schrank, F. A., Mather, N., & McGrew, K. S. (2014). Woodcock-Johnson IV tests of achievement. Rolling Meadows, IL: Riverside.